CLINICAL TRIAL: NCT00004161
Title: A Randomized, Double Blind, Placebo-Controlled Phase II Clinical Trial of N(4-Hydroxy-phenyl)Retinamide (Fenretinide, 4HPR) in Oral Leukoplakia
Brief Title: Fenretinide in Treating Patients With Leukoplakia of the Mouth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CDR0000067401; UAB-9713; NCI-G99-1626
Record Dates: First submitted 1999-12-10; First posted 2004-06-04 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Head and Neck Cancer
Keywords: lip and oral cavity cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Mouth Neoplasms | interventions — Fenretinide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral fenretinide daily (except days 1-3 each month) for 6 months. Patients then receive oral fenretinide daily (except days 1-3 each month) for 6 months. Patients are followed every 3 months.
  Interventions: Drug: fenretinide
- Arm II (Experimental): Patients receive oral placebo daily (except days 1-3 each month) for 6 months. Patients then receive oral fenretinide daily (except days 1-3 each month) for 6 months. Patients are followed every 3 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: fenretinide
  Arms: Arm I
Drug: Placebo
  Arms: Arm II

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development of or treat early cancer. Fenretinide may be an effective drug in treating leukoplakia.

PURPOSE: Randomized phase II trial to study the effectiveness of fenretinide in treating patients who have leukoplakia of the mouth.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine modulation by fenretinide of surrogate endpoint markers of oral mucosal carcinogenesis in patients with oral dysplastic leukoplakia. II. Determine whether fenretinide will cause significant modulation of intermediate endpoint markers and significant regression of oral dysplastic leukoplakia in this patient population. III. Compare the ability of fenretinide and placebo to modulate surrogate endpoint biomarkers in this patient population. IV. Document the degree of recurrence of oral dysplastic leukoplakia after the administration of fenretinide, both at the same site and at new sites.

OUTLINE: This is a randomized, double blind, placebo controlled study. Patients are randomized to 1 of 2 treatment arms: Arm I: Patients receive oral fenretinide daily (except days 1-3 each month) for 6 months. Arm II: Patients receive oral placebo daily (except days 1-3 each month) for 6 months. Patients then receive oral fenretinide daily (except days 1-3 each month) for 6 months. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven dysplastic leukoplakia greater than 1 cm in diameter

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 Platelet count at least 125,000/mm3 Hemoglobin at least 12.0 g/dL Hepatic: Bilirubin less than 1.5 mg/dL SGOT less than 2 times upper limit of normal (ULN) Renal: Creatinine less than 1.7 mg/dL Cardiovascular: No symptomatic coronary artery disease No uncontrolled hypertension No prior coronary artery bypass No acute myocardial infarction in the past year Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective barrier contraception for 1 month prior, during, and for 12 months after study Fasting serum triglyceride less than 2 times ULN Cholesterol less than 350 mg/dL No hypersensitivity to vitamin A or retinoids No active malignancy No concurrent acute or chronic medical or psychiatric condition that would preclude compliance or toxicity assessment No concurrent and severe night blindness

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: At least 3 months since prior chronic high dose (greater than 30,000 IU/day) vitamin A (retinol) At least 1 month since other prior retinoids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1997-06; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Determine modulation by fenretinide of surrogate endpoint markers of oral mucosal carcinogenesis in patients with oral dysplastic leukoplakia. | baseline to 6 months

SECONDARY OUTCOMES:
Determine whether fenretinide will cause significant modulation of intermediate endpoint markers and significant regression of oral dysplastic leukoplakia in this patient population. | baseline to 6 months
Compare the ability of fenretinide and placebo to modulate surrogate endpoint biomarkers in this patient population. | baseline to 6 months
Document the degree of recurrence of oral dysplastic leukoplakia after the administration of fenretinide, both at the same site and at new sites. | baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Samuel W. Beenken, MD, Study Chair — University of Alabama at Birmingham
Locations (1):
- University of Alabama Comprehensive Cancer Center, Birmingham, Alabama, United States